CLINICAL TRIAL: NCT04340869
Title: The Effect of Using Two Desensitizing Agents Alone and In Combination on Dentin Permeability and Hypersensitivity
Brief Title: Treatment of Dentin Hypersensitivity Using Different Desensitizing Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, ebtsam kassab, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC18-145
Record Dates: First submitted 2020-03-02; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Theobromine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Theobromine (Experimental): Natural extract from Cocoa
  Interventions: Other: Theobromine
- Remin Pro (Active Comparator): Fluoride , Hydroxyapatite , and Xylitol
  Interventions: Other: Remin Pro
- Combination (Experimental): Remin Pro and Theobromine
  Interventions: Other: Theobromine; Other: Remin Pro

INTERVENTIONS:
Other: Theobromine — Natural extract from Cocoa
  Arms: Combination; Theobromine
Other: Remin Pro — Remin Pro
  Arms: Combination; Remin Pro

SUMMARY:
Treatment of Dentin Hypersensitivity Using Theobromine , Remin Pro , and Combination of Both Materials

ELIGIBILITY:
Inclusion Criteria:

* Patients that aged 18-50 years.
* Patients in good general health.
* Patients that have accessible teeth demonstrating signs of sensitivity.

Exclusion Criteria:

* • Any chronic debilitating disease that could influence study outcomes.

  * Partial dentures, orthodontic appliances, implants or restorations in a poor state of repair that could influence study outcomes.
  * Intolerance or hypersensitivity to the study desensitizing agents or their ingredients.
  * Desensitising treatment or tooth bleaching within 8 weeks of screening.
  * Daily use of medications that might influence the perception of pain.(

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale pain score | 1 month
  0 = no pain to 10=severe exagerated pain

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University , Faculty of Dental medicine for Girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes